CLINICAL TRIAL: NCT05892367
Title: Transbrachial Access for Interventions in Patients With Peripheral Arterial Occlusive Disease: Evaluation of Local Complications With or Without Post-interventional Immobilization of the Upper Extremity
Brief Title: Transbrachial Access for Interventions in Patients With Peripheral Arterial Occlusive Disease
Acronym: TBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wilhelminenspital Vienna (Other)
Responsible Party: Principal Investigator, Edda Skrinjar, M.D., M.D., Wilhelminenspital Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TBA 1.2
Record Dates: First submitted 2018-02-04; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Complication of Treatment
Keywords: transbrachial access, intervention, bleeding, hematoma
MeSH Terms: conditions — Hemorrhage; Hematoma | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Control group: compression bandage Study group: compression bandage and positioning splint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Application of a compression bandage following transbrachial puncture for 24 hours
  Interventions: Other: Transbrachial Access for Interventions
- Study group (Active Comparator): Application of a compression bandage and a positioning splint following transbrachial puncture for 24 hours
  Interventions: Other: Transbrachial Access for Interventions

INTERVENTIONS:
Other: Transbrachial Access for Interventions — Adding a positioning splint in addition to compression bandage after intervention in order to guarantee immobilization of puncture site

SUMMARY:
The aim of the present study is an evaluation, whether an immobilization of the upper extremity by means of a positioning splint can help to reduce the incidence of local complications after transbrachial puncture for peripheral arterial interventions, or not.

DETAILED DESCRIPTION:
Increasing numbers of peripheral arterial interventions are performed via transbrachial access leading to a higher number of local complications at the puncture site. Patients are demonstrating complications, such as hematoma, false aneurysm, secondary hemorrhage and arterial stenosis or occlusion.

Due to not standardized post-interventional procedure regarding to immobilization a higher risk for local puncture site complication can occur. Usually, a compression bandage its applied to the brachial puncture site. Within this randomized study, patients randomized to the study group will receive an additional splint for 24 hours to ensure an immobilization of the affected arm.

Following the removal of the compression dressing, and the splint in the study group, a duplex ultrasound its performed in order to detect local alterations and pathologies of the brachial artery.

This examination is repeated for each patient in the course of an outpatient control six weeks post-interventionally. Pathologies are documented and treated if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients suffering from peripheral arterial occlusive disease with indicated interventions via an transbrachial access (puncture of the left or right brachial artery)
* age > 18 years
* approval to participate

Exclusion Criteria:

* unability or refusal to participate
* dialysis patients/AV-fistula interventions
* usage of closure devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of local complications at the puncture site | 6 weeks
  Local complications as hematoma, bleeding, pseudoaneurysm, arterial dissection, arterial stenosis, arterial occlusion, AV fistula detected by ultrasound 24 hours after intervention and at time of follow-up six weeks after treatment

SECONDARY OUTCOMES:
Post-interventional pain at puncture site | 24 hours
  Evaluation of local pain according to V.A.S. score by asking patients after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Assadian, Prim. PD Dr., Principal Investigator — Vascular and Endovascular Surgery, Klinik Ottakring
Locations (1):
- Department of Vascular and Endovascular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No